CLINICAL TRIAL: NCT04300894
Title: "Mamma Mia" for Perinatal Health and Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HM20017197; 1R01HD100395 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Usual care group (No Intervention): Usual prenatal and postpartum care involves regular visits with one's health care provider while pregnant and after the baby is born.
- Mamma Mia group (Experimental): Usual prenatal/postpartum care plus use of the "Mamma Mia" program
  Interventions: Device: Mamma Mia
- Mamma Mia Plus group (Experimental): Usual prenatal/postpartum care plus use of the "Mamma Mia" program plus occasional contacts from study staff
  Interventions: Device: Mamma Mia; Other: Mamma Mia Plus

INTERVENTIONS:
Device: Mamma Mia — Users of the Mamma Mia program progress through the intervention in a sequence of modules.
  Every day that a module should be completed, you will receive a notification with a reminder to access the program. By clicking on the reminder, you can access that particular day's session content. Modules involve a variety of information and activities; for example, there are guided mindfulness practices, information on breastfeeding, instructional videos on how to interpret your baby's cries, and discussions on how to have effective discussions with your partner or healthcare provider about your needs.
  Arms: Mamma Mia Plus group; Mamma Mia group
Other: Mamma Mia Plus — Participants will use the Mamma Mia program, plus receive contact (phone calls or emails or texts) from study staff every few months.
  Arms: Mamma Mia Plus group

SUMMARY:
The purpose of this research study is to find out about ways to enhance well-being during pregnancy and the postpartum period (after the baby is born). The "Mamma Mia" program and/or guided support from study staff ("Mamma Mia Plus") may be helpful because the app provides skills and information related to many important topics during and after pregnancy. This study will allow us to learn more about whether and how the program is helpful to women.

DETAILED DESCRIPTION:
This study will compare findings in women who do not use the program ("usual care group") versus women who use the program ("Mamma Mia group") versus women who use the program and receive regular contact from study staff ("Mamma Mia Plus"). The study will assess well-being, depression, stress, and anxiety as well as whether certain factors (for example, women's age, type of healthcare provider, amount of social support) are related to the effects of the program. For women randomized to use the program, the study will also collect information about the time spent using it and the modules completed.

Usual prenatal and postpartum care involves regular visits with participant's women's health care provider while pregnant and after the baby is born. In this study, participants will receive continue receiving usual care. In addition, participants will be randomly assigned (like the flip of a coin) to participate in one of the following groups:

1. The "usual care group", or
2. The "Mamma Mia group" (which is to use the "Mamma Mia" program regularly), or
3. The "Mamma Mia Plus group" (which is to use the program regularly plus receive regular contact with study staff).

There is a 1 chance in 3 of being assigned to each of the three groups. participants have an equal chance of being assigned to any one of the groups.

Participants in the "usual care group" will be asked to do the following things:

1. Complete survey questions at entrance into the study.
2. Complete survey questions every few months (see schedule below).

Participants in the "Mamma Mia group" will be asked to do the following things:

1. Complete survey questions at entrance into the study.
2. Use the "Mamma Mia" program on a regular basis (on average: weekly for about 10 minutes) from entering study until six months postpartum; participants will receive an email reminder to complete modules when they should be completed.
3. Complete survey questions every few months.

Participants in the "Mamma Mia Plus group" will be asked to do the following things:

1. Complete survey questions at entrance into the study.
2. Use the "Mamma Mia" program on a regular basis (on average: weekly for about 10 minutes) from entrance into the study until six months postpartum.
3. Complete survey questions every few months.
4. Participants will receive phone calls or emails or texts (depending upon participant preference) from study staff every few months.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman <25 weeks gestation;
* age 18 or older;
* speak, read, and understand English;
* have the ability to access an internet/mobile-based program (via computer, tablet, or smartphone), and have a working phone number and a working email address.

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1953 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in depression symptom severity | Baseline to 6 months postpartum, about 11 months
  measured by the Edinburgh Postpartum Depression Scale

SECONDARY OUTCOMES:
Change in subjective well-being | Baseline to 6 months postpartum, about 11 months
  Measured using Satisfaction with Life Scale
Change in anxiety | Baseline to 6 months postpartum, about 11 months
  Measured by the State-Trait Anxiety Scale
Change in stress | Baseline to 6 months postpartum, about 11 months
  Measured by the Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Kinser, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinser PA, Moyer S, Jones HA, Jallo N, Popoola A, Thacker L, Russell S, Olavesen ES, Sundrehagen T, Hare MM, Xia B, Garthus-Niegel S, Haga S, Drozd F. Perceptions of the Mamma Mia program, an internet-based prevention strategy for perinatal depression symptoms. PLOS Ment Health. 2025 Apr 3;2(4):e0000138. doi: 10.1371/journal.pmen.0000138. eCollection 2025. PMID 41661763

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04300894/ICF_000.pdf